CLINICAL TRIAL: NCT05276869
Title: Is Arabic Version of WeeFIM Instrument Reliable and Feasible Enough to Measure Functional Independence in Egyptian Children With Burns?
Brief Title: Reliability and Feasibility of WeeFIM Instrument to Measure Functional Independence in Pediatric Burns
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Mohamed othman, professor, Cairo University
Other Study IDs: 012/003578
Record Dates: First submitted 2022-02-28; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Burns
Keywords: WeeFIM instrument; functional independence; pediatric burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: from 3 to 7 years included 36 patients
  Interventions: Other: WeeFIM instrument
- group B: from 8 to 16 years included 17 patients
  Interventions: Other: WeeFIM instrument

INTERVENTIONS:
Other: WeeFIM instrument — In a formative setting, the WeeFIM tool examines functional independence in kids aged 6 months to 7 years old. It can also be used with children over the age of 7 who show functional ability. The instrument may be controlled by observational data or a meeting, and it takes 15 to 20 minutes to create [10].

SUMMARY:
PURPOSE:

Is to test the feasibility and the reliability of the Arabic version of wee functional independence measure (weeFIM) in children with healed burns.

BACKGROUND:

Since kids are the most influenced casualty of burn and they may have lasting disabilities because of this harm, consequently they should have care in evaluation and treatment procedure in exploration.

There are two main instruments that can be utilized to evaluate the function of young kid's which are the Functional independence measure for kids (WeeFIM) instrument and the Pediatric evaluation of disability inventory (PEDI) instrument.

Therefore, the aim of this study was to investigate the reliability and feasibility of the Arabic version of the WeeFIM instrument in kids from 3 years to 16 years of age with healed burn.

HYPOTHESES:

Arabic version of WeeFIM questionnaire will not be feasible and reliable to measure and report the functional outcome of kids with healed burns.

RESEARCH QUESTION:

Is the Arabic version of weeFIM instrument feasible and reliable enough to measure and report the functional outcome of children with healed burns?

DETAILED DESCRIPTION:
1. First the weeFIM will undergo forward Arabic translation followed by English backward translation.
2. Second the instrument will be adapted to Egyptian accent.
3. Third the process of filling of questionnaire will be applied. It will be either parent filled or child filled. And will be performed by interview for illiterate patients.
4. Last, statistical analysis for feasibility and reliability will be performed.

ELIGIBILITY:
Inclusion Criteria:

* patients who had a healed burn with an age from 3 years to 16 years.
* All participants or their parents had to be able to read, write, and speak Arabic
* They had passed two weeks post-burn.

Exclusion Criteria:

* Children with a history of neurological impairment or orthopedic surgery to the limbs or spine.
* those with severe burns (4th degree burns), extensive burn is >60%.
* infected burn wounds.
* other medical conditions that might impair physical performance.
* children with any medical illness present in the previous month.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Enrollment of participants was done for all children who meet the inclusion criteria. The demographic details about each parent and child were noted, and screening was done for adherence to inclusion and exclusion criteria. The tool was given to all children aged 3 years to 16 years who were hospitalized in one of the two places for more than two weeks after the burn.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2021-09-05 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Reliability | Change from Baseline, after 2 weeks postburn.
  The reliability of the Arabic version of the WeeFIM instrument was assessed by a test-retest procedure. First, the researcher collected a random sample of participants. Second, the researchers explained the procedure to the participants. Third, the researchers explained the items of the questionnaire to the participants. Fourth, the participants were asked to fill the scale with score-1. Fifth, one week apart, they were asked to re-fill the scale with score-2. Sixth, test-retest reliability was analysed by using Pearson Correlation Coefficient (PCC) and internal consistency was measured by using Cronbach's alpha Coefficient.
Content validity | Change from Baseline, after 2 weeks postburn.
  In this study, content validity (items' relevance and adequacy for the intended use) of the Arabic version of the WeeFIM instrument was assessed. Content validity deals with the extent to which an instrument reflects the meaningful elements of the content without extraneous elements [19].

CONTACTS AND LOCATIONS:
Overall Officials: eman othman, PhD, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in bee venom or ulcer . we will share the results of this study within 1 year following publication.
Supporting Information: SAP, ICF
Time Frame: 1 year after publication
Access Criteria: the criteria will be assessed by the publication of the trial in an international journals.